CLINICAL TRIAL: NCT07312474
Title: Epidemiological, Clinical and Biological Characteristics of Human Anaplasmosis Cases in Alsace: a Retrospective and Multicenter Study
Brief Title: Epidemiological, Clinical and Biological Characteristics of Human Anaplasmosis Cases in Alsace
Acronym: ANARETRO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9458
Record Dates: First submitted 2025-12-11; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Human Anaplasmosis
Keywords: Human Anaplasmosis; Ticks; Tick bite; Severe cytopenias; Respiratory distress syndrome; Septic shock; Neurological disorders; Macrophage activation syndrome
MeSH Terms: conditions — Anaplasmosis; Tick Bites; Cytopenia; Respiratory Distress Syndrome; Shock, Septic; Nervous System Diseases; Macrophage Activation Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anaplasmosis is a bacterial infection caused by the intracellular bacterium Anaplasma phagocytophilum and transmitted by ticks. This bacterium is present in approximately 1% of ticks in Alsace. This infection is responsible for clinical manifestations that are most often mild, including fever, headache, and myalgia, occurring 2 to 3 weeks after a tick bite. However, this infection can be accompanied by potentially serious or even fatal complications, including severe cytopenias, acute respiratory distress syndrome, septic shock, severe neurological disorders, hemorrhagic manifestations, macrophage activation syndrome, and multiple organ failure. Mortality is variable and appears to be higher in American studies, where it is around 4%. Treatment is well-established and relies on doxycycline, which is highly effective. Although a few cases have been described in France, these are mostly isolated cases or short series of cases, whereas Belgium, Poland, and Slovenia have reported numerous cases. Thus, there is a lack of data on French cases, and given that Alsace is in a region with a high prevalence of tick-borne diseases, data is needed to better understand the epidemiology and to better identify suspected cases in order to provide appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjct (≥18 years)
* Presenting with a PCR-confirmed infection of Anaplasma

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subjct (≥18 years) having a PCR-confirmed infection of Anaplasma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Mortality of cases of human anaplasmosis in Alsace | Up to 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France